CLINICAL TRIAL: NCT02761213
Title: Efficacy of Reduced Volume Oral Sulfate Solution (SUPREP) Compared With PEG Plus Ascorbic Acid for Screening Colonoscopy: Single Center, Single Blinded Prospective Randomized Study
Brief Title: Oral Sulfate Solution (SUPREP) Versus Polyethylene Glycol (PEG) Plus Ascorbic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bo-In Lee (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Bo-In Lee, MD, PhD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KC16MISV0004
Record Dates: First submitted 2016-04-22; First posted 2016-05-04 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Cathartic Colon

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral sulfate solution (OSS) (Experimental): oral sulfate solution (OSS)
  Interventions: Drug: Oral sulfate solution (OSS)
- 2-L PEG/Asc (Active Comparator): low-dose polyethylene glycol plus ascorbic acid (2-L PEG/Asc)
  Interventions: Drug: 2-L PEG/Asc

INTERVENTIONS:
Drug: Oral sulfate solution (OSS) — Oral sulfate solution (OSS)
  Other Names: SUPREP
  Arms: Oral sulfate solution (OSS)
Drug: 2-L PEG/Asc — Low-dose polyethylene glycol plus ascorbic acid (2-L PEG/Asc) COOLPREP is a proprietary name of 2-L PEG/Asc.
  Other Names: COOLPREP
  Arms: 2-L PEG/Asc

SUMMARY:
The aims of the present study is to compare oral sulfate solution (OSS) with low-dose polyethylene glycol plus ascorbic acid (2-L PEG/Asc) for bowel cleansing efficacy.

DETAILED DESCRIPTION:
High-quality bowel cleansing is critical to effective colonoscopy. Studies in the past decade have demonstrated that many clinical practices continue to have rates of adequate preparation as low as 60% to 80%.

Low-volume preparations for colonoscopy are designed to improve patient tolerability, another important aspect of bowel preparation. In addition, low-volume preparations should ideally not sacrifice efficacy. There are few data comparing the efficacy of available low-volume bowel preparations.

In this study, we describe a prospective, single-blind, randomized, controlled trial comparing oral sulfate solution (OSS) (SUPREP, Braintree Laboratories, Braintree, Mass) with low-dose polyethylene glycol plus ascorbic acid (2-L PEG/Asc).

ELIGIBILITY:
Inclusion Criteria:

* people who receive colonoscopy
* aged : 18-80
* people who sign the consent

Exclusion Criteria:

* those aged over 80 years
* the disabled
* intestinal obstruction
* severe constipation
* previous history of bowel resection
* liver cirrhosis
* heart failure or ischemic heart disease within 6 months
* inflammatory bowel disease
* pregnant women
* severe renal insufficiency
* people who refuse to sign the consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BPPS) | during colonoscopy
Aronchick scale | during colonoscopy
  Aronchick scale is a commonly used bowel preparation scale to grade the adequacy of cleansing of colonic segments or the entire colon.

SECONDARY OUTCOMES:
Tolerability by a patient questionnaire using 5-point Likert scale | on arrival at the endoscopy unit before colonoscopy
  to assess tolerability of each bowel preparation
Safety by measuring hemodynamic and biochemical data | at baseline (in the clinic be- fore booking the colonoscopy) and on arrival at the en- doscopy suite
  Biochemical data will be measured only in case of necessity such as weakness, mental change or numbness.
Colonoscopic finding: whether there is erythematous mucosal change or apthous ulcers | during colonoscopy
Percentage of cecal intubation | during colonoscopy
Insertion time | during colonoscopy
Withdrawal time | during colonoscopy
Adenoma detection rate | during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Bo-In Lee, MD, PhD, Study Director — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM; ASGE/ACG Taskforce on Quality in Endoscopy. Quality indicators for colonoscopy. Am J Gastroenterol. 2006 Apr;101(4):873-85. doi: 10.1111/j.1572-0241.2006.00673.x. No abstract available. PMID 16635231
- [Background] Bannas P, Bakke J, Patrick JL, Pickhardt PJ. Automated volumetric analysis for comparison of oral sulfate solution (SUPREP) with established cathartic agents at CT colonography. Abdom Imaging. 2015 Jan;40(1):11-8. doi: 10.1007/s00261-014-0186-x. PMID 24965898
- [Background] Rex DK, DiPalma JA, McGowan J, Cleveland Mv. A comparison of oral sulfate solution with sodium picosulfate: magnesium citrate in split doses as bowel preparation for colonoscopy. Gastrointest Endosc. 2014 Dec;80(6):1113-23. doi: 10.1016/j.gie.2014.05.329. Epub 2014 Jul 12. PMID 25028274
- [Derived] Lee HH, Lim CH, Kim JS, Cho YK, Lee BI, Cho YS, Lee IS, Choi MG. Comparison Between an Oral Sulfate Solution and a 2 L of Polyethylene Glycol/Ascorbic Acid as a Split Dose Bowel Preparation for Colonoscopy. J Clin Gastroenterol. 2019 Nov/Dec;53(10):e431-e437. doi: 10.1097/MCG.0000000000001137. PMID 30308546